CLINICAL TRIAL: NCT06847997
Title: Videoconferencing for the Management of Paediatric Dyspnoea in an Emergency Medical Call Centre: the VISIODYS-PED Randomised Controlled Study Protocol
Brief Title: Videoconferencing for the Management of Paediatric Dyspnoea in an Emergency Medical Call Centre
Acronym: VISIODYS-PED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VISIODYS-PED
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-03

CONDITIONS: Out-of-hospital Setting; Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard medical dispatching process (Control group) (No Intervention): The emergency physician dispatcher conducts a standard medical dispatching process.
- Addition of telemedicine to standard medical dispatching process (Experimental Group) (Experimental): The emergency physician dispatcher conducts a standard medical dispatching process with the addition of telemedicine using video calls.
  Interventions: Other: Addition of telemedicine to standard medical dispatching process (Experimental Group)

INTERVENTIONS:
Other: Addition of telemedicine to standard medical dispatching process (Experimental Group) — In the experimental group, the same approach is used, with the addition of telemedicine using video calls. Callers are invited to use their smartphone camera to enable real-time video assessment. The medical dispatcher sends a secure link (via a platform provided by Enovacom, Nomadeec, Bordeaux, France) to the caller's smartphone, allowing video streaming through a secure internet connection. Once the link is validated by the caller, the live video feed from the smartphone camera is transmitted directly to the dispatcher's computer screen, providing a visual evaluation to support clinical decision-making.
  Arms: Addition of telemedicine to standard medical dispatching process (Experimental Group)

SUMMARY:
Dyspnoea is defined as the sensation of difficult or uncomfortable breathing experienced by a patient. It is a significant concern in emergency care, accounting for 8% of calls to the emergency medical call centre (EMCC) and 10% of Emergency department (ED) admissions. Among paediatric patients, dyspnoea accounts from 14-27% of ED admissions, exhibiting notable seasonal variation. Approximately 10% of these patients require hospitalisation, and 1-3% of cases progress to respiratory failure. All these patients require a comprehensive clinical examination to accurately identify signs of severity, ensuring the timely initiation of specialized and effective treatment.

In France, patients are encouraged to contact the local EMCC before visiting an ED. Medical dispatchers assess the clinical condition by phone, based on medical history, symptoms and current treatment. Based on this assessment, the medical dispatcher determines the appropriate decision which may include providing medical advice, directing the patient to an ED, or deploying a mobile intensive care unit (MICU). Seven percent of calls to an EMCC involve paediatric cases, with nearly half concerning children under six years of age with hyperthermia and dyspnoea as most complaints, particularly during epidemic periods. The medical assessment of paediatric dyspnoea by EMCC is particularly challenging. The inability of children to articulate their symptoms, coupled with parents difficulty in describing the situation - often exacerbated by anxiety - creates significant obstacles. Furthermore, the absence of a direct observation by the physician adds to the complexity and could lead to an inappropriate triage and management.

Telemedicine uses communication technologies for remote consultations, electronic record management, and document sharing. It enables real-time visual evaluation, thereby improving diagnostic accuracy and decision-making. While evidence supports its benefits in managing adult dyspnoeic patients, further research is essential to validate its efficacy in paediatric settings, particularly within EMCC.

This study will aim to evaluate the effectiveness of telemedicine within an EMCC and utilising real-time visualization in reducing inappropriate triage of children requiring care for acute dyspnoea.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3 months to 5 years
* Call from parent(s) to an EMCC for dyspnea or shortness of breath or difficulty breathing as main complaint
* Parent or witness with a phone/tablet equipped with a camera
* Emergency consent or oral consent given by the holder(s) of parental authority to the physician dispatcher

Exclusion Criteria:

* Child in life-saving emergency
* Known absence of a telephone network required for the use of video calls
* Call made by an individual who does not hold parental authority
* Communication difficulties with the holder(s) of parental authority, not allowing for a clear and fair information
* Person not benefiting from a social security scheme or through a third party
* Child who has already participated in the study

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 339 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients inaccurately managed | 24 hours
  The primary endpoint is the proportion of patients inaccurately managed (over-triage or under-triage)
  Over-triage is defined as a situation where a patient is:
  1. Directed to an ED following the call, but does not require any specific treatment, diagnostic tests, or hospitalisation, within 24h following the primary call, or
  2. Managed by the deployment of a MICU, despite not requiring specific treatment or transfer to an ED, within 24h following the primary call.
  Under-triage is defined as a situation where a patient is kept at home with medical advice or directed to a family practitioner after the primary call AND later dispatched to hospital by a family practitioner or after a second call to an EMCC for dyspnoea, or hospitalised or dead within 24h following the primary call.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Marjanovic, MD PhD, Principal Investigator — Poitiers University Hospital; Erwan Ripley, MD, Principal Investigator — Poitiers University Hospital
Locations (1):
- CHU Poitiers, Poitiers, France, France

IPD SHARING:
Plan to Share IPD: Undecided